CLINICAL TRIAL: NCT02533596
Title: Elimination of Cardiac and Inflammatory Biomarkers and Adipokines by Therapeutic Plasma Exchange
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: TPE-5343-2010
Record Dates: First submitted 2015-02-27; First posted 2015-08-27 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-02

CONDITIONS: Antibody-mediated Rejection; Autoimmune Reaction Mediated by Immune Complex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * blood samples
  * plasma samples from TPE waste bag
Oversight: Data Monitoring Committee: No

SUMMARY:
Therapeutic plasma exchange (TPE) is an established treatment modality for the acute removal of pathophysiological relevant mediators in various diseases. Adipokines have recently been found to play an important role in a variety of immunologic diseases. However, in many of these disease states cardiac and inflammatory involvement is common and biomarkers are routinely used for diagnosis or assessment of therapeutic success. The effect of TPE on biomarkers used in the clinical routine has not been investigated. The aim of this study is to determine adipokine and cardiac biomarker removal during TPE therapy.

DETAILED DESCRIPTION:
We performed a observational prospective single-centered study. Every patient received two consecutive therapeutic plasma exchange (TPE) sessions during the study. Plasma exchange therapy was performed using either the Spectra Optia® or the Octo Nova® apheresis system. Anticoagulation was applied either by heparin or citrate. The prescribed dose of exchange volume of every TPE treatment was 1.1-times the individual calculated total plasma volume, using the Nadler-Allen equation. A substitute fluid with 5% albumin concentration was used in every treatment. Blood samples for measurement of different adipokines (resistin, leptin, soluble ICAM-1, soluble CD40 ligand, monocyte chemoattractant protein-1 (MCP-1), soluble tumor necrosis factor receptor (sTNF-R) as well as cardiac and inflammatory biomarkers and routine chemistry were drawn before (pre-TPE) and at the end (post-TPE) of the first and second TPE session.

ELIGIBILITY:
Inclusion Criteria:

* indication for TPE
* age between 18 and 80 years
* written informed consent

Exclusion Criteria:

* need for fresh-frozen plasma as replacement fluid
* participation in another study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary hospital patients after kidney transplantation with humoral rejection and patients with other antibody mediated diseases.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Percentage decrease in serum levels of C-reactive protein by TPE | Up to five days after enrollment
  Elimination of C-reactive protein by TPE measured by the decrease in serum levels after two consecutive TPE sessions.
Percentage decrease in serum levels of Troponin T by TPE | Up to five days after enrollment
  Elimination of cardiac biomarkers Troponin T by TPE measured by the decrease in serum levels after two consecutive TPE sessions.
Percentage decrease in serum levels of procalcitonin by TPE | Up to five days after enrollment
  Elimination of procalcitonin by TPE measured by the decrease in serum
Percentage decrease in serum levels of NT-proBNP by TPE | Up to five days after enrollment
  Elimination of NT-proBNP by TPE measured

SECONDARY OUTCOMES:
Percentage decrease in serum levels of adipokines by TPE | Up to five days after enrollment
  Elimination of adipokines by TPE measured by the decrease in serum levels after two consecutive TPE sessions.
Total eliminated amount of Troponin T by TPE | Up to five days after enrollment
  Elimination of Troponin T by TPE measured by the total eliminated amount in the exchanged plasma.
Total eliminated amount of NT-proBNP by TPE | Up to five days after enrollment
  Elimination of NT-proBNP by TPE measured by the total eliminated amount in the exchanged plasma.
Total eliminated amount of procalcitonin by TPE | Up to five days after enrollment
  Elimination of procalcitonin by TPE measured by the total eliminated amount in the exchanged plasma.
Total eliminated amount of C-reactive protein by TPE | Up to five days after enrollment
  Elimination of C-reactive protein by TPE measured by the total eliminated amount in the exchanged plasma.
Total eliminated amount of adipokines by TPE | Up to five days after enrollment
  Elimination of adipokines by TPE measured by the total eliminated amount in the exchanged plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Jan T Kielstein, Prof., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany